CLINICAL TRIAL: NCT01406548
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dose Study to Assess the Safety and Efficacy of Multiple Dosing Regimens of BPS804 in Post Menopausal Women With Low Bone Mineral Density
Brief Title: Safety and Efficacy of Multiple Dosing Regimens of BPS804 in Post Menopausal Women With Low Bone Mineral Density
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Mereo BioPharma (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBPS804A2203
Record Dates: First submitted 2011-07-11; First posted 2011-08-01 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Osteopenia; Osteoporosis
Keywords: Osteopenia; osteoporosis; low bone mineral density
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — setrusumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- BPS804 dosing frequency 1 (Experimental): Subjects dosed 20mg/Kg BPS804 monthly
  Interventions: Drug: BPS804 20mg/Kg
- placebo dosing frequency 1 (Placebo Comparator): Subjects dosed with matching placebo to 20mg/Kg BPS804 monthly
  Interventions: Drug: Placebo to 20mg/Kg BPS804
- BPS804 dosing frequency 2 (Experimental): Subjects dosed with 20mg/Kg BPS804 quarterly
  Interventions: Drug: BPS804 20mg/Kg
- placebo dosing frequency 2 (Placebo Comparator): Subjects dosed with matching placebo to 20mg/Kg BPS804 every 3 months
  Interventions: Drug: Placebo to 20mg/Kg BPS804
- BPS804 dosing frequency 3 (Experimental): Subjects dosed with 20mg/Kg BPS804 weekly
  Interventions: Drug: BPS804 20mg/Kg
- Placebo dosing frequency 3 (Placebo Comparator): Subjects dosed with matching placebo to 20mg/Kg BPS804 weekly
  Interventions: Drug: Placebo to 20mg/Kg BPS804

INTERVENTIONS:
Drug: BPS804 20mg/Kg
  Arms: BPS804 dosing frequency 1; BPS804 dosing frequency 2; BPS804 dosing frequency 3
Drug: Placebo to 20mg/Kg BPS804
  Arms: Placebo dosing frequency 3; placebo dosing frequency 1; placebo dosing frequency 2

SUMMARY:
This study is designed to provide information on the safety, tolerability, pharmacokinetics (PK) and bone biomarker response following multiple BPS804 administration in multiple dosing regimens. This information will permit a comparison of the possible risks and benefits of different dosing regimens of the study drug to enable optimal doses and dose intervals to be tested in subsequent studies.

DETAILED DESCRIPTION:
This study was conducted and previously posted by Novartis. The record was transferred to Ultragenyx in February 2021.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (natural or surgically induced menopause)
* Low bone mineral density (BMD), as defined by a T score or equivalent BMD absolute value (g/cm2) for lumbar spine of between -2.0 and -3.5, inclusive
* Body mass index (BMI) must be within the range of 18 to 35kg/m2. Subjects must weigh between 45 and 120kg inclusive to participate.
* 25-(OH) vitamin D serum level of ≥ 15ng/ml
* Serum calcium within normal limits

Exclusion Criteria:

* Subjects with suspected neural foraminal stenosis (e.g., cervical, spinal, lumbar), or history of Bell's palsy, cranial nerve disorders, temporomandibular joint and muscle disorders.
* Subjects who have an increased baseline risk of osteosarcoma: Paget's disease of the bone or unexplained and clinically significant elevations of alkaline phosphatase and/or subjects who have received radiation therapy involving the skeleton.
* Subjects with any known bone diseases other than postmenopausal osteoporosis.
* Subjects with a history of an osteoporotic fracture (e.g., vertebral fracture, fragility fracture of the wrist, radius, humerus, hip, or pelvis).
* Subjects who are regularly using or have regularly used agents affecting bone metabolism:

  * Calcitonin, estrogen, SERMs (raloxifene, Tamoxifen, etc.), Tibolone progestin, or androgens within the last three (3) months prior to screening.
  * Any oral bisphosphonate, lithium chloride, fluoride or systemic glucocorticosteroids (p.o. or i.v.) where the total dose exceeds 750 mg of prednisone or equivalent within the last year prior to screening.
  * Any previous use of denusomab (ProliaTM), parathyroid hormone (ForteoTM), and/or PTH analogs, strontium ranelate, or parenteral formulations of bisphosphonates.
* Current disease(s) known to influence calcium metabolism including hyperparathyroidism, hypoparathyroidism, hypocalcemia or hypercalcemia.
* Any disease, abnormality or deformation of the spine (e.g., scoliosis, ankylosing spondylitis, osteophytes) or hip (e.g., joint prosthesis) which would preclude the proper acquisition of a lumbar spine DXA (L1-L4) or femur DXA, respectively.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline to month 9 in bone mineral density at the lumbar spine for the individual BPS804 groups and pooled placebo arms. | 9 months
The number (percent) of subjects experiencing adverse events or serious adverse events | 9 months

SECONDARY OUTCOMES:
Change from baseline during 9 months of serological bone biomarkers for the individual BPS804 groups and pooled placebo arms. | 9 months
Characterization of the PK profile of BPS804: area under the plasma concentration-time curve (AUC) | 260 days
Characterization of the PK profile of BPS804: time to reach the maximum Characterization of the PK profile of BPS804: maximum plasma concentration (Cmax) | 260 days
Characterization of the PK profile: time to reach the maximum concentration (Tmax) | 260 days
Characterization of the PK profile of BPS804: half-life (T1/2) | 260 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (4):
- United States (4):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Berlin, New Jersey
  - Novartis Investigative Site, Duncansville, Pennsylvania